CLINICAL TRIAL: NCT04273659
Title: Combining Cereals With Pulses - Reduced Gastrointestinal Symptoms?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Kaisa Linderborg, Professor of Molecular Food Sciences (acting), University of Turku
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Pulses
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Unidentified Gastrointestinal Symptoms Following Pulses Consumption
MeSH Terms: interventions — Pulse; Edible Grain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulses and Cereal 1 (Experimental): Pulses and cereal 1 containing study product is served. Dietary intervention.
  Interventions: Dietary Supplement: Pulses and cereals
- Pulses and Cereal 2 (Experimental): Pulses and cereal 2 containing study product is served. Dietary intervention.
  Interventions: Dietary Supplement: Pulses and cereals

INTERVENTIONS:
Dietary Supplement: Pulses and cereals — Dietary intervention. Ingestion of pulses with cereals and gastrointestinal health.

SUMMARY:
The aim of the study is to compare self-reported gastrointestinal symptoms and intestinal fermentation rates of the study products as measured by breath hydrogen and methane in adult population with self-reported mild abdominal sensitivity to pulses. The study products are a pulse products with two different cereals.

DETAILED DESCRIPTION:
The study is a randomized, controlled, double-blind, cross-over intervention trial. The aim is to recruit 25 subjects to the trial. The study will be conducted with a cross-over setting, where the subjects will go through exposure meals and breath gas measurement two times (two different test products) in a randomized order. The study meals are identical in appearance but differ in fiber content. After study breakfast the breath gases are analyzed every 15 minutes during 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with subjective experience of gut symptoms after consumption of pulses
* Celiac disease and wheat allergy excluded by antigen test
* Age 18-65
* BMI 18,5 - 30
* Normal liver, thyroid and kidney functions

Exclusion Criteria:

* Celiac disease, Crohn's disease, ulcerative colitis or acute diverticulitis
* Any medication affecting the gastrointestinal tract (e.g. laxatives and acid-suppressive drugs)
* Antibiotic treatment within previous 3 months
* Blood donation or participation to another clinical trial within one month prior to study entry

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Breath gases | Day 4
  Breath hydrogen and methane are measured by Gastrocheck device.

SECONDARY OUTCOMES:
Gastrointestinal symptoms (self-reported) | Day 1-4
  Gastrointestinal symptoms as measured as questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa Linderborg, PhD, Principal Investigator — Department of Biochemistry, University of Turku
Locations (1):
- Department of Biochemistry, University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided